CLINICAL TRIAL: NCT02191852
Title: A Pharmacokinetic Study on the Antioxidant Activity of Seresis® in the Skin: an Open, Uncontrolled, Non-randomized Intra-individual Pilot Trial in Healthy, Young Female Volunteers
Brief Title: Pharmacokinetic Study of Seresis® in the Skin in Healthy Young Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1135.4
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (1):
- Seresis® (Experimental): 2 capsules per day for a period of 16 consecutive weeks
  Interventions: Drug: Seresis®

INTERVENTIONS:
Drug: Seresis®

SUMMARY:
Study to evaluate the total antioxidant capacity of Seresis® (with Thiobarbituric acid reactive substances (TBARS) assays)) in the skin; as well as in buccal mucosa cells (BMCs) and in plasma, compared to baseline values; furthermore to detect the quantitative enrichment of individual antioxidant compounds contained in the product and to investigate whether or not some of them accumulate in target tissues such as skin, BMCs and plasma

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers between 18 and 30 years
* With skin type II or skin type III
* BMI < 25
* Non-smokers
* Volunteers who have given their written informed consent according to Good Clinical Practice (GCP) and local regulations

Exclusion Criteria:

* Any serious disorder that may interfere with her participation to the trial and evaluation of the safety of the test drug (e.g. liver and/or renal disease, hypervitaminosis A, psychic disorder, etc.), and/or treatment with chronic medication
* Pre-treatment (less than 2 weeks prior to inclusion in this trial) and/or concomitant treatment with any drug that may influence the trial symptomatology and may interfere with evaluation of the safety of the test drug (e.g. vitamins and minerals supplementation)
* Relevant allergy or known hypersensitivity to the investigational drug or its excipients
* High performance sports
* Alcohol and drug abuse according to Diagnostic and Statistics Manual, Version IV (DSM-IV)
* Female volunteers in child-bearing age not using adequate means of birth control (contraceptive pills, Intrauterine devices (IUDs), sterilisation)
* Pregnancy and/or lactation
* Known abnormal values of the lab tests (if detected after enrolment, subjects will continue the treatment provided there are no medical objections)
* Abnormal values of low density lipoproteins (LDL) and triglycerides (TGL) levels in blood
* Participation in another clinical trial within the last 4 weeks and concurrent participation in another clinical trial
* Specific dietary requirements that do not allow the volunteers to meet the dietary guidelines set out for this study

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 1999-06; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Total antioxidant capacity in skin biopsies | Day 0, Day 112

SECONDARY OUTCOMES:
Total antioxidant capacity in skin biopsies | Day 0, Day 56
Total antioxidant capacity in buccal mucosa cells (BMCs) | Day 0, 14, 28, 42, 56, 84, 112
Total antioxidant capacity in plasma | Day 0, 14, 28, 42, 56, 84, 112
Plasma levels of vitamin C and E and carotenoids | Day 0, 14, 28, 42, 56, 84, 112
Levels of vitamin E and carotenoids in skin biopsies | Day 0, 56, 112
Levels of vitamin E and carotenoids in BMCs | Day 0, 14, 28, 42, 56, 84, 112
Number of subjects with adverse events | up to 119 days
Assessment of tolerability by investigator on a 4-point scale | Day 112
Assessment of tolerability by volunteers on a 4-point scale | Day 112
Number of patients with abnormal changes in laboratory parameters | up to 112 days